CLINICAL TRIAL: NCT05297292
Title: A Multicenter, Randomized, Double-blind, Positive-controlled, Seamless Design Phase II/III Clinical Study to Evaluate the Efficacy and Safety of Recombinant Anti-VEGF Humanized Monoclonal Antibody Injection (Code MW02) in the Treatment of Neovascular (Wet) Age-related Macular Degeneration (nAMD)
Brief Title: A Study to Evaluate the Efficacy and Safety of MW02 in the Treatment of nAMD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW02-2020-CP301
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lucentis-0.5mg（Q4w） (Active Comparator): It is administered once every 4 weeks for 48 weeks. Intravitreal injection was used, and the dose was 0.5mg.
  Interventions: Drug: Lucentis
- MW02-1.0mg（Q4w） (Experimental): It is administered once every 4 weeks for 48 weeks. Intravitreal injection was used, and the dose was 1.0mg.
  Interventions: Drug: MW02
- MW02-1.5mg（Q4w） (Experimental): It is administered once every 4 weeks for 48 weeks. Intravitreal injection was used, and the dose was 1.5mg.
  Interventions: Drug: MW02
- MW02（Q8w） (Experimental): It is administered once every 4 weeks for 3 consecutive times, and then once every 8 weeks for 48 weeks.
  Interventions: Drug: MW02

INTERVENTIONS:
Drug: MW02 — MW02 is a recombinant anti-VEGF humanized monoclonal antibody injection.
  Arms: MW02-1.0mg（Q4w）; MW02-1.5mg（Q4w）; MW02（Q8w）
Drug: Lucentis — a recombinant anti-VEGF humanized monoclonal antibody injection
  Other Names: ranibizumab
  Arms: Lucentis-0.5mg（Q4w）

SUMMARY:
The purpose of this study is to compare the efficacy and safety of MW02 versus Lucentis in the treatment of neovascular age-related macular degeneration.The study was divided into two stages. The first stage was to explore the dose and the second stage was to explore the frequency of administration.

ELIGIBILITY:
Main Inclusion Criteria:

1. fully understand this research and sign ICF; Willing to follow and be able to complete all study procedures;
2. Age ≥ 50 years old, < 80 years old, male or female;
3. Active CNV lesions in fovea and/or parafovea secondary to nAMD , which have not been treated in the study eye 3 months before screening;
4. The BCVA of the study eye is 73~24 letters (including boundary value), which is equivalent to 20/40 to 20/320 of Snellen's visual acuity chart.
5. CNV area of the study eye≥50% of the total lesion area.

Main Exclusion Criteria:

1. There is subretinal or intraretinal hemorrhage in the study eye, and the bleeding area is ≥ 50% of the total lesion area, or it is located in the fovea and the area is ≥ 1 optic disc area;
2. The study eye has scar, fibrosis, geographic atrophy and dense hard exudation under the fovea.
3. CNV caused by non-nAMD exists in the study eye (such as trauma, pathological myopia, multifocal choroiditis, ocular histoplasmosis, vascular stripes, etc.);
4. The study eye has any eye diseases or medical history other than nAMD that may affect central vision and/or macular examine (diabetic retinopathy, retinal vein occlusion, retinal detachment, macular hole, macular epiretinal membrane, retinal pigment epithelium tear involving macular, vitreous macular traction syndrome, optic nerve disease, etc.);
5. Intravitreous hemorrhage occurred in the study eye within 30 days before the first administration.
6. The study eye has received the following intraocular surgery within 90 days, or has previously received various macular laser treatments (such as macular transposition, transpupillary thermotherapy, macular photocoagulation, vitrectomy, optic nerve incision, optic nerve sheath incision, etc.) (except those who have received Vitepofin-photodynamic therapy, cataract surgery and YAG posterior capsulotomy more than 3 months before screening) or have performed external eye surgery within 30 days;
7. The study eye has used corticosteroids in the eye or in the whole body within 3 months or injected corticosteroids around the globe within 30 days before the first administration;
8. The study eye has poorly controlled glaucoma (defined as intraocular pressure≥25 mmHg after anti-glaucoma treatment), and/or has received glaucoma filtering surgery (such as trabeculectomy, scleral bite, non-penetrating trabecular surgery, etc.);
9. The study eye has high myopia with diopter≥8D
10. The study eye has refractive interstitial turbidity and/or myosis that affect fundus or OCT examination;
11. Aphakia (except intraocular lens) or rupture of posterior capsule of lens (except YAG laser posterior capsulotomy after intraocular lens implantation more than 30 days before the first administration);
12. Scleromalacia exists in the study eye.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Best Corrected Visual Acuity (BCVA) | At week 52
  Change from Baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study(ETDRS) letter score at week 52.

SECONDARY OUTCOMES:
Change from Baseline in BCVA | baseline to week 52
  Change from Baseline in BCVA as measured by ETDRS letter score over the study duration.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China